CLINICAL TRIAL: NCT02509819
Title: The Influence of Heel Wedge Properties on Roll-over of the Intrepid Dynamic Exoskeletal Orthosis (IDEO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrea J. Ikeda, Research Prosthetist, Brooke Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2015.017d
Record Dates: First submitted 2015-07-27; First posted 2015-07-28 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Physical Disability
Keywords: rehabilitation; IDEO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Military Performance Lab testing (Experimental): Subjects who use IDEOs will come to the Military Performance Lab for one test session during which they will walk in standardized shoes with six different foam heel wedges (Heel Cushion Material Bulk (foam) from Kingsley Manufacturing Company) in random order. Control data will also be collected on able-bodied individuals. Control subjects will also come to the MPL for one test session in which they will walk using the same standardized shoes. For all subjects, biomechanical gait data will be collected as the subjects walk along a walkway in the MPL. This data will be used to calculate roll-over shape, instantaneous radius of curvature, COP velocity, and ankle moment.
  Interventions: Device: Heel Cushion Material Bulk (foam)

INTERVENTIONS:
Device: Heel Cushion Material Bulk (foam) — The heel wedge is made of a rubber style urethane foam. Heel wedges of specified heights and durometers will be inserted into the standard shoes, one at a time, during the test session only. The heel wedges used during the test session are made of the same foam as the heel wedges that are used clinically.

SUMMARY:
The Intrepid Dynamic Exoskeletal Orthosis (IDEO) is a type of ankle foot orthosis designed to reduce pain and improve function for individuals with foot/ankle pain and/or weakness. Because the IDEO restricts ankle movement, the geometry and mechanics of the device must be designed to allow for a smooth roll-over as the patient walks with the IDEO. The heel wedge, while not physically part of the IDEO, is an integral part of the IDEO-heel wedge-shoe "system". The goal of this research is to determine how heel wedge properties may contribute to the smoothness of roll-over during gait. Insight into the effects of heel wedge properties on roll-over will help optimize the design of the IDEO-heel wedge-shoe "system" and may produce guidelines for the customization of these features.

DETAILED DESCRIPTION:
The proposed study includes a between groups comparison (for Aim 1) and a fully repeated crossover design (for Aim 2). It will be conducted in the Military Performance Lab (MPL) at the Center for the Intrepid (CFI), Brooke Army Medical Center, Joint Base San Antonio (JBSA)Fort Sam Houston, Texas. Subjects who use IDEOs will come to the Military Performance Lab for one test session during which they will walk in standardized shoes with six different heel wedges in random order. Control data will also be collected on able-bodied individuals. Control subjects will also come to the MPL for one test session in which they will walk using the same standardized shoes. For all subjects, biomechanical gait data will be collected as the subjects walk along a walkway in the MPL. This data will be used to calculate roll-over shape, instantaneous radius of curvature, Center of Pressure (COP) velocity, and ankle moment.

ELIGIBILITY:
IDEO Group

Inclusion Criteria:

* DEERS (Defense Enrollment Eligibility Reporting System) eligible patients at the CFI
* 18 - 55 years old
* Have a unilateral lower extremity injury resulting in foot/ankle weakness and/or pain
* Currently using an IDEO
* Use of the IDEO for greater than two weeks
* Able to ambulate without an assistive device
* Able to comply with gait analysis
* Able to provide written informed consent

Exclusion Criteria:

* Neurologic, musculoskeletal or other disease state affecting the contralateral limb that limits normal locomotion
* Spinal cord injury or central nervous system pathology
* Medical or psychological disease that would preclude safe gait analysis (ex. severe traumatic brain injury, stroke, renal failure, heart disease, severe anemia, etc.)
* Pain level of 4 or greater on a 0-10 scale
* Any open wound or infection on the foot
* Pregnancy

Control Group

Inclusion Criteria:

* DEERS eligible
* 18 - 55 years old
* Have no lower extremity injury which affects normal locomotion
* Able to comply with gait analysis
* Able to provide written informed consent

Control Group Exclusion Criteria:

* Neurologic, musculoskeletal or other disease state that limits normal locomotion
* Previous lower extremity injury requiring surgery (e.g. anterior cruciate ligament tear, femur fracture, etc) or currently affecting normal locomotion
* Any pain that affects normal locomotion
* Any open wound or infection on the foot
* Spinal cord injury or central nervous system pathology
* Medical or psychological disease that would preclude safe gait analysis (ex. severe traumatic brain injury, stroke, renal failure, heart disease, severe anemia, etc.)
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04-25 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
Roll-over shape | 2 hours
  This will be calculated by determining the COP location in the coordinate system of the shank. The shape will be described by the calculated arc length and best-fit radius of curvature
Instantaneous radius of curvature | 2 hours
  This will be calculated by taking the derivative of the anterior-posterior progression of the COP with respect to the shank angle
COP velocity | 2 hours
  This will be calculated by taking the derivative of the COP anterior-posterior position
Ankle moment | 2 hours
  This will be calculated from the Ground Reaction Force (GRF) vector relative to the ankle joint center

CONTACTS AND LOCATIONS:
Overall Officials: Andrea J Ikeda, MS, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States